CLINICAL TRIAL: NCT04752176
Title: Evaluation of the Elimination of Tinnitus and Hyperacusis by the ØREBLUE® Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mayfair Developments (Industry)
Responsible Party: Sponsor
Other Study IDs: MAY001-PMCF001
Record Dates: First submitted 2021-02-03; First posted 2021-02-12 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Tinnitus; Hyperacusis
Keywords: Tinnitus; hyperacusis; Medical device; ØREBLUE® Method
MeSH Terms: conditions — Tinnitus; Hyperacusis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tinnitus group: At least 20 patients suffering from tinnitus will be enrolled in the study.
  Interventions: Device: ØREBLUE® Method
- Hyperacusis group: At least 20 patients suffering from hyperacusis will be enrolled in the study.
  Interventions: Device: ØREBLUE® Method

INTERVENTIONS:
Device: ØREBLUE® Method — The ØREBLUE® Method combines 2 inseparable therapeutic approaches that will be personalized, one dedicated to the auditory symptom (personalized sound therapy based on music and delivered through a helmet as part of the device), the other dedicated to the psychology of the subject.
  Sound rehabilitation will be based on successive treatment sequences. The 1st sequence includes 30 hours of listening, at a rate of 2 hours / day, 5 days a week. A period of 4 to 6 weeks is necessary before carrying out a new sequence. The second sequence (and subsequent ones when necessary, respecting a 4-to-6-weeks window in between) of sound rehabilitation consists of 20 hours distributed as for the first sequence.

SUMMARY:
Tinnitus and hyperacusis are two hearing disorders that can severely impact the patient and their quality of life, as they may induce sleeping disorders, concentration troubles, social life disturbances. Mayfair Developments has created and developed the innovating ØREBLUE® method in order to relieve, possibly completely, tinnitus and hyperacusis symptoms. The ØREBLUE® method relies on a medical device, CE marked, that consists of an auditory stimulation box associated with five softwares. This medical device diffuses thanks to a headphone a specific and personalized sound therapy treatment for the patient. This retrospective, observational study aims at collecting data about the ØREBLUE® method used in routine care and describing its efficacy on tinnitus and hyperacusis.

DETAILED DESCRIPTION:
Tinnitus is a clinical symptom indicative of abnormal stimulation of the auditory system characterized by the perception of chronic sound in the absence of an external sound source and that only the affected subject perceives intrusively.Its presence can occur independently unilaterally, bilaterally, or be described as perceived in the center of the head and can be heard continuously or intermittently at varying levels of intensity and frequency. There are two types of tinnitus depending on whether it can be detected with a stethoscope by the doctor (objective tinnitus) or only heard by the subject (subjective tinnitus). Many consequences, such as anxiety, depression and sleep disorders, linked to suffering from tinnitus will impact daily life in different forms.

Both types of tinnitus may be accompanied by a higher intolerance to noise which is called hyperacusis.Hyperacusis is defined as an intolerance (and not a finer sensitivity to sounds) to environmental sound levels, the intensity of which, of varying intensity, represents neither risk nor inconvenience for people with normal hearing, but which induces discomfort or pain in people with hyperacusis.

In these clinical situations, the ØREBLUE® method is an innovative treatment with the objective of eliminating the symptoms of tinnitus and hyperacusis depending on the group to which the subject belongs. Its innovative character is based on the design of a sound signal processing device, CE marked as medical device, developed by Mayfair Developments. This technological innovation has been developed to respond specifically to the hearing profile of each subject and to provide personalized rehabilitation of their hearing sphere.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years old
* Subject seen in consultation in the investigational site from CE marking up to 2 years thereafter,
* Sufficient ENT investigations,
* Satisfactory general condition: non-invalidating medical history (ENT disorders and others),
* The subject agrees to work on the emotional part linked to their condition,
* Permanent and disabling tinnitus and/or hyperacusis, with the following characteristics for tinnitus: subjective, chronic (present for more than 1 year), resistant to usual treatments (medication, hearing aid with or without masking, psychotherapy) continued for a minimum of 6 months, severe tinnitus, disabling tinnitus (measurement with numerical scale score and THI questionnaire),
* Patient informed about the study and has no objection to take part

Exclusion Criteria:

* Proven presence of an anxiety disorder of claustrophobia type,
* History of neurological disease, in particular personal or family history of epilepsy or seizure (infantile hyperthermic convulsions, or other type of seizure),
* Serious psychiatric history or attempted autolysis, concomitant use of antidepressant and neuroleptic treatment,
* Bilateral cophosis,
* Medication monitoring that can generate more or less tinnitus,
* More than 6 months since the end of the last treatment or therapy against tinnitus,
* For women: possibility of pregnancy (absence of effective contraception or certain menopause), breastfeeding woman,
* Context of medico-legal litigation and / or concomitant participation in another protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be retrospectively collected from consecutive patients suffering from tinnitus and/or hyperacusis and treated in the investigational site by the ØREBLUE® Method since the CE marking date and up to 3 years-time.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in Discomfort | From baseline through study completion, an average of 10 months.
  Discomfort level is rated on a numerical scale, from 0 to 10, where 0 means "no discomfort" and 10 means "indescribable discomfort".

SECONDARY OUTCOMES:
Hyperacusis Symptoms change | From baseline through study completion, an average of 10 months.
  Hyperacusis symptoms are assessed with the Hyperacusis Handicap Inventory (HHI) questionnaire
Hyperacusis discomfort level | From baseline through study completion, an average of 10 months.
  Disconfort level due to hyperacusis, in Decibels, during audiometric measurements
Tinnitus Symptoms change | From baseline through study completion, an average of 10 months.
  Tinnitus symptoms are assessed with the Tinnitus Handicap Inventory (THI) questionnaire
Quality of life change | From baseline through study completion, an average of 10 months.
  Quality of life is assessed through WHODAS 2.0 questionnaire
Sleep quality change | From baseline through study completion, an average of 10 months.
  Sleep quality is assessed through the Pittsburgh Sleep Quality Index (PSQI)
Depression | From baseline through study completion, an average of 10 months.
  Depression is assessed through the Beck Depression Inventory (BPI) questionnaire
Anxiety | From baseline through study completion, an average of 10 months.
  Anxiety is assessed through the State-Trait Anxiety Inventory (STAI) questionnaire
Anxiety level | From baseline through study completion, an average of 10 months.
  Anxiety level is rated on a numerical scale, from 0 to 10, where 0 means "no anxiety" and 10 means "worst anxiety".
Appetite level | From baseline through study completion, an average of 10 months.
  Appetite level is rated on a numerical scale, from 0 to 10, where 0 means "no impact on appetite" and 10 means "worst impact on appetite".
Energy level | From baseline through study completion, an average of 10 months.
  Energy level is rated on a numerical scale, from 0 to 10, where 0 means "no impact on energy" and 10 means "worst impact on energy".
Emotionality | From baseline through study completion, an average of 10 months.
  Emotionality is rated on a numerical scale, from 0 to 10, where 0 means "no impact on emotionality" and 10 means "worst impact on emotionality".
Concentration ability | From baseline through study completion, an average of 10 months.
  Concentration ability is rated on a numerical scale, from 0 to 10, where 0 means "no impact on concentration ability" and 10 means "worst impact on concentration ability".
Hopelessness feeling | From baseline through study completion, an average of 10 months.
  Hopelessness feeling is rated on a numerical scale, from 0 to 10, where 0 means "no hopelessness feeling" and 10 means "worst hopelessness feeling".
Isolation feeling | From baseline through study completion, an average of 10 months.
  Isolation feeling is rated on a numerical scale, from 0 to 10, where 0 means "no isolation feeling" and 10 means "worst isolation feeling".

CONTACTS AND LOCATIONS:
Overall Officials: Natacha CHETRITT-BONNEYRAT, Principal Investigator — Mayfair Developments
Locations (1):
- Hearing Institute of Resources, La Rochelle, France